CLINICAL TRIAL: NCT06762132
Title: A Clinical Study to Explore the Safety and Efficacy of CD33 CAR-T Cell in Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024025
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: CD33 CAR-T
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CD33 CAR T-cells

INTERVENTIONS:
Biological: CD33 CAR T-cells — Each subject receive CD33 CAR T-cells by intravenous infusion
  Other Names: CD33 CAR T-cells injection

SUMMARY:
A Clinical Study on the Safety and Effectiveness of targeting CD33 CAR-T Cell in the treatment of Relapsed/Refractory Acute Myeloid Leukemia

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety and efficacy of CD33 CAR-T Cell in patients with relapsed or refractory acute myeloid leukemia. It is planned to enroll 15-27 participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, age ≥ 18 years old;
* 2. CAR-T cells can be prepared normally, or who have failed to prepare autologous CAR-T cells (including the number of autologous lymphocytes <1×10^9 or the expansion during the preparation process is insufficient or cannot reinfusion);
* 3. Patients diagnosed with CD33 positive acute myeloid leukemia (AML) through histological or immunological examination，and CD33 positive expression rate >80%;
* 4. Complies with the 2016 WHO classification for AML diagnosis and meets the diagnostic criteria for recurrence and refractory acute myeloid leukemia in the "Chinese Guidelines for the Diagnosis and Treatment of relapsed and refractory acute myeloid leukemia (2017 edition)", and currently there are no clinically relevant treatments or suitable clinical trials for registration:
* a) Diagnostic criteria for recurrent AML: After complete remission (CR), leukemia cells reappear in peripheral blood or primitive cells in bone marrow>0.050 (excluding other reasons such as bone marrow regeneration after consolidation chemotherapy) or leukemia cell infiltration appears outside the bone marrow;
* b) Diagnostic criteria for refractory AML: initial treatment cases that have failed to respond to two courses of standard protocol treatment; Patients who relapse within 12 months after consolidation and intensive treatment after CR; Patients who relapse after 12 months but fail conventional chemotherapy; Patients with 2 or more relapses; Persistent extramedullary leukemia;
* 5. The number of primitive cells (promyelocytes and/or promyelocytes) in the bone marrow > 5% (morphology) and/or > 1% (flow cytometry detection);
* 6. Total bilirubin ≤ 51 μmol / L, ALT and AST ≤ 3 times of the upper limit of normal value, serum creatinine ≤ 176.8 μmol / L；
* 7. Echocardiography shows left ventricular ejection fraction (LVEF) ≥ 50%;
* 8. There is no active pulmonary infection, and the oxygen saturation during air inhalation is more than 92%;
* 9. The estimated survival time is more than 3 months;
* 10. ECOG score was 0-2;
* 11. Pregnant/lactating women, or male or female patients who have fertility and are willing to take effective contraceptive measures at least 6 months after the last cell infusion during the study period;
* 12. Those who voluntarily participated in this trial and provided informed consent;

Exclusion Criteria:

* 1. Patients with the history of epilepsy or other CNS disease;
* 2. Patients with prolonged QT interval time or severe heart disease;
* 3. Active infection with no cure;
* 4. Active infection of hepatitis B virus or C virus ;
* 5. Before using any gene therapy products;
* 6. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 7. Suffering from other uncontrolled diseases that the researchers consider unsuitable for joining;
* 8. Infected with AIDS virus;
* 9. Any situation that researchers believe may increase the risk to the subjects or interfere with the trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Complete response (CR), and complete response with incomplete hematologic recovery (CRi) | Up to 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Duration of remission ,DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Overall survival, OS | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause
Leukemia-Free Survival, LFS | Up to 2 years after Treatment
  The time from CAR-T infusion torecurrence or metastasis

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China